CLINICAL TRIAL: NCT07047131
Title: A Resorbable Versus a Non-resorbable Bone Substitute at Immediate Post-extractive Single Implants Immediately Loaded: a Multicentre Randomised Controlled Trial
Brief Title: Resorbable vs Non-resorbable Bone Substitute at Immediate Post-extractive Single Implants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Marco Esposito (Network)
Responsible Party: Sponsor-Investigator, Marco Esposito, Associate Professor, Marco Esposito
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2301201902319
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Tooth Extraction; Bone Graft; Alveolar Bone Loss; Dental Implant
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resorbable Bone Substitute (GTO®) (Experimental): Patients receive a fully resorbable bone substitute (GTO®) to fill the gap between the implant and the buccal bone wall during immediate post-extraction implant placement.
  Interventions: Biological: GTO® (fully resorbable bone substitute)
- Partially Resorbable Bone Substitute (Apatos®) (Active Comparator): Patients receive a partially resorbable bone substitute (Apatos®) to fill the gap between the implant and the buccal bone wall during immediate post-extraction implant placement.
  Interventions: Biological: Apatos® (partially resorbable bone substitute)

INTERVENTIONS:
Biological: GTO® (fully resorbable bone substitute) — Collagenated heterologous cortico-cancellous porcine bone mix + thermogelling copolymer with collagen (GTO®, OsteoBiol®, Tecnoss®)
  Arms: Resorbable Bone Substitute (GTO®)
Biological: Apatos® (partially resorbable bone substitute) — Porcine cortical bone granules (Apatos Cortical®, OsteoBiol®, Tecnoss®) stabilized with TSV Gel®, a thermogelling copolymer with collagen.
  Arms: Partially Resorbable Bone Substitute (Apatos®)

SUMMARY:
This study compares two bone graft materials used when placing a dental implant right after tooth removal. One graft fully dissolves (GTO®), the other only partly (Apatos®).

The goal is to see which one better preserves bone and improves appearance around the implant.

DETAILED DESCRIPTION:
This multicenter, double-blind randomized controlled trial aims to compare the clinical, radiographic, and aesthetic outcomes of two xenogeneic bone substitutes, GTO® (fully resorbable) and Apatos® (partially resorbable), used in post-extractive sockets at the time of immediate implant placement.

Eligible patients are adults requiring a single-tooth extraction in the maxilla or mandible, followed by immediate implant placement.

The primary outcome is peri-implant bone volume changes over time, assessed using CBCT scans.

Secondary outcomes include implant and crown failure, implant stability, marginal bone level changes on periapical radiographs, and aesthetic outcomes evaluated using the pink esthetic score based on clinical photographs.

Patients will be followed up to 5 years after loading.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring at least one single immediate post-extractive implant.
* At least 18 year old, able to understand and to sign an informed consent
* There must be sufficient bone to allow the placement of at least a 3.5 mm diameter and 8.5 mm long implant.
* After tooth extraction there must be a potential gap of at least 2 mm from the buccal inner bone plate and the implant surface.

Exclusion Criteria:

* General contraindications to implant surgery.
* Immunosuppressed or immunocompromised patients.
* Patients irradiated in the head and/or neck.
* Uncontrolled diabetes.
* Pregnancy or lactation.
* Active periodontal disease
* Poor oral hygiene and motivation.
* Addiction to alcohol or drugs.
* Psychiatric problems and/or unrealistic expectations
* Patients with an acute infection (abscess) in the site intended for implant placement.
* Patients unable to commit to a 5-year follow-up.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* patients referred only for implant placement if follow-ups cannot be done at treatment centre.
* Patients participating in other studies, if the present protocol could not be fully adhered to. In case of doubts please contact the study coordinator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2030-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in peri-implant bone volumes | From enrollment to 5 years after implant loading
  Volumetric changes in peri-implant tissues will be measured using limited-view CBCT scans taken at implant placement (baseline), 1 year, and 5 years after loading. The main endpoint is the difference in bone volume between baseline and 1 year.

SECONDARY OUTCOMES:
Number of participants with crown or implant failure | From enrollment to 5 years after implant loading
  Defined as the inability to place the crown due to implant failure, or the need for crown replacement for any reason. Implant failure is defined as implant mobility and/or any infection dictating implant removal and any mechanical complications rendering the implant unusable (e.g. implant fracture). The stability of each individual implant will be measured by the blinded outcome assessor manually by assessing the stability of the crown using the handles of two metallic instruments at 1 and 5 years after loading.
Number of biological and biomechanical complications | From enrollment to 5 years after implant loading
  Biological and biomechanical complications will be recorded and reported by study group. Examples of biological complications are: fistula, peri-implantitis. Examples of biomechanical complications are fracture of the metal screws, loosening of the crown, fracture of the ceramic lining.
Peri-implant marginal bone level changes | From enrollment to 5 years after implant loading
  Periapical digital radiographs will be made with the paralleling technique at implant placement, at 1 and 5 years of loading. In case of an unreadable radiograph, the radiograph must be made again. Peri-implant marginal bone levels will be measured using the Image J (National Institutes of Health, Bethesda, Maryland, USA) software. The software will be calibrated for every single image using the known implant length or, if the full implants is not visible on the radiograph, the implant diameter. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured at both mesial and distal sides and averaged. Bone level at single implants will be averaged at group level.
Aesthetic evaluation using the Pink Esthetic Score (0-14; higher scores = better outcome) | From enrollment to 5 years after implant loading
  Aesthetic evaluation of the clinical pictures taken at delivery of the final crown (baseline), at 1- and 5-year follow-ups, on a computer screen by an independent blinded dentist. The pictures of the vestibular and occlusal aspects must include the two adjacent teeth. The aesthetic evaluation will be done following thePink Esthetic Score, a validated index that ranges from 0 (worst aesthetic outcome) to 14 (best aesthetic outcome), based on soft tissue parameters around the implant implant-supported crown.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Esposito, Dentistry, Principal Investigator — Associate Professor
Locations (1):
- King Juan Carlos University, Madrid, Madrid, Spain

REFERENCES:
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Thalmair T, Fickl S, Schneider D, Hinze M, Wachtel H. Dimensional alterations of extraction sites after different alveolar ridge preservation techniques - a volumetric study. J Clin Periodontol. 2013 Jul;40(7):721-7. doi: 10.1111/jcpe.12111. Epub 2013 May 5. PMID 23647007
- [Background] De Angelis N, Felice P, Pellegrino G, Camurati A, Gambino P, Esposito M. Guided bone regeneration with and without a bone substitute at single post-extractive implants: 1-year post-loading results from a pragmatic multicentre randomised controlled trial. Eur J Oral Implantol. 2011 Winter;4(4):313-25. PMID 22282729
- [Background] Esposito M, Grusovin MG, Polyzos IP, Felice P, Worthington HV. Interventions for replacing missing teeth: dental implants in fresh extraction sockets (immediate, immediate-delayed and delayed implants). Cochrane Database Syst Rev. 2010 Sep 8;2010(9):CD005968. doi: 10.1002/14651858.CD005968.pub3. PMID 20824846

DOCUMENTS (1):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT07047131/Prot_000.pdf